CLINICAL TRIAL: NCT07128979
Title: Efficacy and Safety Evaluation of Ruscus Aculeatus L in Patients With Hemorrhoids: A Randomized, Double-blind Phase IV Clinical Trial
Brief Title: Efficacy and Safety Evaluation of Ruscus Aculeatus L in Patients With Hemorrhoids
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Collaborators: Atabay Kimya Sanayi Ticaret A.S. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KAEK-18
Record Dates: First submitted 2025-08-07; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Hemorrhoid
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group: Neoven 225 mg capsules (Active Comparator): Patients in this group will only use Neoven 225 mg capsules orally. There will be no signs or inscriptions on the capsules regarding their contents. The duration of the study is determined as 42 days. A total of 378 mg of total ruscogenin (ruscogenin/neoruscogenin mixture obtained by extraction method) will be taken orally using one Neoven capsule orally with meals twice a day. A total of 84 capsules will be given to the patients.
  Interventions: Drug: Neoven 225 mg capsules
- Control group (Placebo Comparator): Patients in this group will only receive an oral placebo capsule designed for this study. There will be no signs or inscriptions on the capsules regarding their contents. The duration of the study is determined as 42 days. During this period, one placebo capsule will be taken orally twice a day with meals. A total of 84 capsules will be given to the patients, and their use will be questioned by phone on the 7th and 14th days of the treatment and the number of uses will be checked at the end of the treatment. Failure to use all of the capsules will be considered as a criterion for exclusion from the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neoven 225 mg capsules — Patients in this group will only use Neoven 225 mg capsules orally. There will be no signs or inscriptions on the capsules regarding their contents. The duration of the study is determined as 42 days. A total of 378 mg of total ruscogenin (ruscogenin/neoruscogenin mixture obtained by extraction method) will be taken orally using one Neoven capsule orally with meals twice a day. A total of 84 capsules will be given to the patients, and their use will be questioned by phone on the 7th and 14th days of the treatment and the number of uses will be checked at the end of the treatment. Failure to use all of the capsules will be considered as a criterion for exclusion from the study.
  Arms: Study group: Neoven 225 mg capsules
Drug: Placebo — Patients in this group will only receive an oral placebo capsule designed for this study. There will be no signs or inscriptions on the capsules regarding their contents. The duration of the study is determined as 42 days. During this period, one placebo capsule will be taken orally twice a day with meals. A total of 84 capsules will be given to the patients, and their use will be questioned by phone on the 7th and 14th days of the treatment and the number of uses will be checked at the end of the treatment. Failure to use all of the capsules will be considered as a criterion for exclusion from the study.
  Arms: Control group

SUMMARY:
Hemorrhoidal disease is characterized by distal displacement and deterioration of structural integrity of vascular cushions in the anal canal, which physiologically help defecation and continence. Unlike advanced stage (stage IV) hemorrhoids, which require surgical intervention, various topical agents (gels, ointments, creams), oral venoactive drugs, homeopathic and phytotherapeutic products and nutritional supplements are widely used in stage II and III hemorrhoidal disease. The genus Ruscus (family Asparagaceae) is a group of plants native to the Mediterranean basin, Southern and Western Europe, and Iran, represented by perennial, rhizome-based, and evergreen shrubs. Among the species belonging to this genus, Ruscus aculeatus L. has the widest distribution area. The subsoil parts of the Ruscus plant are rich in steroidal saponins and show vasoconstrictor, diuretic, anti-inflammatory and venotonic effects, especially with ruscogenin and neoruscogenin compounds. Due to these properties, R. aculeatus stands out as a traditional phytotherapy agent that has been used for a long time in chronic venous insufficiency. However, there are no controlled clinical studies in the literature evaluating the efficacy and safety of Ruscus aculeatus L. in hemorrhoidal disease. Therefore, this study was aimed to systematically evaluate the contribution of a phytotherapeutic product containing R. aculeatus to the treatment of stage II-III hemorrhoidal patients and to provide scientific evidence of a new and potentially safe herbal treatment option that can be used in the treatment of hemorrhoids.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the efficacy and safety of Neoven 225 mg capsule containing Ruscus aculeatus L. in individuals with stage II-III hemorrhoidal disease according to the Goligher classification.

Hemorrhoidal disease is characterized by distal displacement and deterioration of structural integrity of vascular cushions in the anal canal, which physiologically help defecation and continence. As a result, venous distension, inflammation, erosion, bleeding and thrombosis may develop in hemorrhoidal tissues.

Clinically, depending on the stage of the disease, symptoms such as bright red rectal bleeding during defecation, discomfort around the anus, itching, fecal incontinence, pain and protrusion may occur. However, uncertainty about the pharmacological treatment of hemorrhoidal disease still remains.

Unlike advanced stage (stage IV) hemorrhoids, which require surgical intervention, various topical agents (gels, ointments, creams), oral venoactive drugs, homeopathic and phytotherapeutic products and nutritional supplements are widely used in stage II and III hemorrhoidal disease. Among oral venoactive drugs, synthetic calcium dobesilate, diosmin-hesperidin combination of natural origin, triterpenes and saponins are the most well-known compounds. The genus Ruscus (family Asparagaceae) is a group of plants native to the Mediterranean basin, Southern and Western Europe, and Iran, represented by perennial, rhizome-based, and evergreen shrubs. Among the species belonging to this genus, Ruscus aculeatus L. has the widest distribution area. The subsoil parts of the Ruscus plant are rich in steroidal saponins and show vasoconstrictor, diuretic, anti-inflammatory and venotonic effects, especially with ruscogenin and neoruscogenin compounds. Due to these properties, R. aculeatus stands out as a traditional phytotherapy agent that has been used for a long time in chronic venous insufficiency.

However, there are no controlled clinical studies in the literature evaluating the efficacy and safety of Ruscus aculeatus L. in hemorrhoidal disease. Therefore, this study was aimed to systematically evaluate the contribution of a phytotherapeutic product containing R. aculeatus to the treatment of stage II-III hemorrhoidal patients and to provide scientific evidence of a new and potentially safe herbal treatment option that can be used in the treatment of hemorrhoids.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18-45 with complaints (symptomatic) consistent with hemorrhoidal disease
2. Patients with Stage II and III hemorrhoids according to the Goligher Hemorrhoid Rating system using physical examination (digital rectal examination, anoscopy/rectoscopy performed within a maximum of four weeks before the examination)
3. Patients who have signed the Informed Consent Form

Exclusion Criteria:

* Patients aged <18 and >45 years
* Stage I and IV hemorrhoids according to the Goligher Hemorrhoid Rating system
* Surgery for hemorrhoids at any time
* Injection treatment for multiple hemorrhoids in the last 3 years
* Perianal sepsis, inflammatory bowel disease, colorectal malignancy, or pre-existing sphincter injury within the last 3 years
* Immunodeficiency
* In addition to hemorrhoids, patients with anal fissures and perianal fistulas detected by simultaneous physical examination or anoscopy/rectoscopy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Life for HSS (Hemorrhoid Severity Score) | At the end of the treatment (42nd day)
  Hemorrhoid Severity Score (HSS) is the total score obtained by the sum of the numerical grades of pruritis, pain, prolapse, bleeding and soiling. All the five components in this classification system are graded into four grades ranging from 0 to 3.

SECONDARY OUTCOMES:
Hemorrhoidal Disease Symptom Score (HHSS) | At the end of the treatment (42nd day)
  The HHSS is a scale that is scored based on five main symptoms: pain, bleeding, itching, fecal incontinence, and prolapse. For the frequency rating of these symptoms, the total score is calculated according to the five-point Liekert classification [Never (score=0), Less than once a month (score=1), Less than once a week (score=2), 1-6 days a week (score=3), Every day/always (score=4)]. The total score ranges from 0 to 20.
Visual Analog Scale (VAS) | At the end of the treatment (42nd day)
  A visual scale with a value range between 0 and 10 will be shown to patients for the VAS pain score, and the they will be asked to rate their current pain as "0"; for no pain and "10"; for unbearable severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Haluk Kerim KARAKULLUKCU, MD, Principal Investigator — Sultan Abdulhamid Training and Research Hospital
Locations (1):
- Sultan Abdulhamid Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouskela E, Cyrino FZ, Marcelon G. Effects of Ruscus extract on the internal diameter of arterioles and venules of the hamster cheek pouch microcirculation. J Cardiovasc Pharmacol. 1993 Aug;22(2):221-4. doi: 10.1097/00005344-199308000-00008. PMID 7692161
- [Background] Masullo M, Pizza C, Piacente S. Ruscus Genus: A Rich Source of Bioactive Steroidal Saponins. Planta Med. 2016 Dec;82(18):1513-1524. doi: 10.1055/s-0042-119728. Epub 2016 Nov 8. PMID 27825178
- [Background] Boyle P, Diehm C, Robertson C. Meta-analysis of clinical trials of Cyclo 3 Fort in the treatment of chronic venous insufficiency. Int Angiol. 2003 Sep;22(3):250-62. PMID 14612852
- [Background] Pompilio G, Nicolaides A, Kakkos SK, Integlia D. Systematic literature review and network Meta-analysis of sulodexide and other drugs in chronic venous disease. Phlebology. 2021 Oct;36(9):695-709. doi: 10.1177/02683555211015020. Epub 2021 May 13. PMID 33983078